CLINICAL TRIAL: NCT07050225
Title: Evaluating the Feasibility and Tolerability of a Digital Cognitive Training Intervention in Adults With ADHD: A Randomized, Placebo-controlled Trial
Brief Title: Evaluating a Digital Cognitive Training Intervention in Adults With ADHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCOG_ADHD
Record Dates: First submitted 2025-06-06; First posted 2025-07-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: ADHD
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Problematic Internet Use; PIU; Cognitive Training Intervention; Executive Functioning; Adult ADHD; ADHD Symptoms; Digital Health; Adjunct Therapy; Hyperactivity; Attention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Cognitive Training (Experimental): Participants randomized to the intervention group will receive 1-hour cognitive training sessions three times weekly for 10 weeks. The digital cognitive training platform will consist of personalized gamified cognitive tasks that target individual cognitive deficits associated with ADHD including attention, impulsivity, working memory, and cognitive flexibility.
  Interventions: Other: Digital Cognitive Training
- Digital Non-cognitive Training Intervention (Placebo Comparator): Participants will use a control gamified computer platform matched for time but lacking cognitive training components. Participants will engage in this activity for 1 hour three times a week for a duration of 10 weeks.
  Interventions: Other: Digital Non-cognitive Training Intervention

INTERVENTIONS:
Other: Digital Cognitive Training — This digital cognitive training program uses gamified tasks in order to enhance cognitive skills in an engaging manner using machine learning AI algorithms to target the intervention to individual cognitive skill deficits. It consists of personalized gamified cognitive tasks that target individual cognitive deficits associated with ADHD including attention, impulsivity, working memory, and cognitive flexibility.
  Arms: Digital Cognitive Training
Other: Digital Non-cognitive Training Intervention — This is a gamified computer platform lacking cognitive training components.
  Arms: Digital Non-cognitive Training Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether a digital cognitive training program can reduce symptoms of ADHD, improve executive functioning, and decrease problematic internet use in adults aged 18-65 with a diagnosis of moderate to severe ADHD. The main questions it aims to answer are:

Can digital cognitive training improve executive function, and ADHD symptoms in adults with ADHD?

Does digital cognitive training reduce problematic internet use in this population?

Researchers will compare the digital cognitive training intervention group to a non-cognitive training digital platform to see if the training leads to greater improvements in cognitive and behavioral outcomes.

Participants will:

Complete an 11-week digital cognitive training program (3, 1-hour sessions/week) or placebo intervention (3, 1-hour sessions/week)

Attend baseline, midpoint, and post-intervention assessments

Participate in weekly check-ins to monitor engagement and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Participants must provide informed consent and agree to comply with study protocols for the duration of the study.
* Participants must be fluent in speaking and reading English and able to complete rating scales and assessments.
* Participants must be adults aged 18-65 years.
* Participants must have a clinical diagnosis of ADHD based on DSM-5 Criteria, as confirmed by the Mini Neuropsychiatric interview.
* Participants being treated with pharmacotherapy must be stable and on a consistent dose for at least 6 weeks prior to study entry.
* Participants must have access to a computer capable of running the cognitive training platform.
* Participants must be comfortable operating a computer and be able to log on to the platform without assistance.

Exclusion Criteria:

* Exclude individuals who meet DSM-5 criteria for psychiatric conditions such as borderline personality disorder, schizophrenia, severe depression, or other psychotic disorders as well as neurological conditions such as epilepsy, dementia, and amnesia, that may interfere with cognitive training.
* Exclude participants with active substance use disorders.
* Exclude participants receiving behavioral therapy or undergoing similar cognitive training programs for ADHD and/or PIU.
* Exclude individuals with severe visual, auditory, or motor impairments that affect the ability to perform the digital cognitive training intervention.
* Exclude participants who are uncomfortable using applications or required technology.
* Exclude participants who have changed their treatment regimen in the last 6 weeks.
* Exclude participants who are not fluent in English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants who prematurely withdraw from the study protocol | From enrollment to the end of treatment at 11 weeks
  Tolerability of the digital cognitive training intervention will be assessed by calculating the number of participants who discontinue participation before completing the full 11-week study protocol. Premature withdrawal will be defined as any participant who discontinues the intervention and/or does not complete post-treatment assessments.
The feasibility of digital cognitive training on ADHD symptoms in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Feasibility will be evaluated based on the number of people who contact the study team, percent of people who contact who are eligible, and percent of eligible participants who enroll. Percent of participants lost to follow-up will be a key determinant of feasibility, as well as number of completers.

SECONDARY OUTCOMES:
The effect of digital cognitive training on ADHD symptoms in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  ADHD symptom severity will be measured via the Barkley Adult ADHD Rating Scale (BAARS-IV). The minimum score on the Barkley ADHD Rating Scale is 0, and the maximum score is 54. The scale consists of 18 items, each rated on a scale of 0 to 3, where 0 indicates the absence of the symptom and 3 indicates a high level of severity.
The effects of digital cognitive training on problematic internet use in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Changes in the severity of problematic internet use will be evaluated via changes in Compulsive Internet Use Scale (CIUS) scores.
The effects of digital cognitive training on visual processing and working memory in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Performance on Trails A and B task will be evaluated.
The effects of digital cognitive training on cognitive flexibility in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Performance on Berg's Card Sorting Task will be evaluated.
The effects of digital cognitive training on working memory in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Performance on N-back Task will be evaluated.
The effects of digital cognitive training on verbal short-term and working memory in adults diagnosed with ADHD of moderate-severe severity | From enrollment to the end of treatment at 11 weeks
  Performance on the Digit Span Test will be evaluated.

OTHER OUTCOMES:
Changes on symptoms of anxiety | From enrollment to the end of treatment at 11 weeks
  The Generalized Anxiety Disorder 7-item (GAD-7), a 7-item questionnaire will be used to screen for the severity of symptoms of anxiety. The Generalized Anxiety Disorder 7-item (GAD-7) scale has a minimum score of 0 and a maximum score of 21. The scale uses a 4-point Likert scale for each of its 7 items, ranging from 0 ("Not at all") to 3 ("Nearly every day"). Higher scores indicate more severe anxiety symptoms.
Changes on symptoms of depression | From enrollment to the end of treatment at 11 weeks
  The Patient Health Questionnaire (PHQ)-9, the major depressive disorder (MDD) module of the full PHQ will be used to measure the severity of depressive symptoms. The PHQ-9 is a widely used tool for assessing depression severity. The minimum possible score on the PHQ-9 is 0, and the maximum is 27. Each of the 9 questions is scored from 0 to 3, with higher scores indicating more severe symptoms.
Changes in quality of life | From enrollment to the end of treatment at 11 weeks
  World Health Organization Quality of Life Brief Version (WHOQOL-BREF) will be used to assess impairment and quality of life. The WHOQOL-BREF (World Health Organization Quality of Life Brief Version) is scored on a 1-5 scale for each of the 26 items. These scores are then transformed to a 0-100 scale. The minimum possible score for each domain is 0, representing the worst possible quality of life, and the maximum is 100, representing the best possible quality of life.